CLINICAL TRIAL: NCT07249320
Title: Observational Cohort Study Evaluating Real-World ABRYSVO Vaccine Effectiveness and Impact Against Medically-Attended RSV-related and All-Cause Outcomes Among Infants Born to Individuals Vaccinated During Pregnancy
Brief Title: Evaluating ABRYSVO Maternal Vaccine Effectiveness Among Infants
Status: Active, not recruiting | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: C3671048
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Respiratory Syncytial Virus (RSV)
Keywords: Lower respiratory tract infections; acute respiratory tract infections; RSV; maternal immunization
MeSH Terms: interventions — abrysvo

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Exposed: Infants whose mother received ABRYSVO vaccine during pregnancy 14 days or more before delivery
  Interventions: Biological: ABRYSVO
- Unexposed: Infants born to mothers who did not receive ABRYSVO during pregnancy will be considered unexposed

INTERVENTIONS:
Biological: ABRYSVO — Participants will receive Pfizer's ABRYSVO vaccine as part of standard of care. Vaccine is not administered in this study.
  Groups: Exposed

SUMMARY:
To generate critical evidence to support vaccine policy and implementation, Pfizer will collaborate with Kaiser Permanente Northern California (KPNC) to study the vaccine effectiveness (VE) of ABRYSVO vaccination during pregnancy in a real-world population. The overall research question of this study is: what is the effectiveness of ABRYSVO vaccination during pregnancy against medically-attended (MA) RSV-associated and all-cause infant outcomes in a large, diverse, real-world population? This study will use a retrospective cohort design and will be conducted within an integrated delivery health care organization using electronic medical record (EMR) data collected during routine standard of care clinical encounters. Study outcomes among infants born to ABRYSVO-vaccinated mothers (exposed group) will be compared with those among infants born to ABRYSVO-unvaccinated mothers (comparison group) initially from birth through 6 months of age, with later assessments from birth through 12 months of age and through 24 months of age as the infants reach these age thresholds and their data become available. There are two categories of outcomes of interest in this study: RSV-specific infant outcomes and non-specific all-cause infant outcomes, assessed within several follow-up windows (birth through 6 months of age, birth through 12 months of age, and/or birth through 24 months of age, depending on the outcome).

Identification of RSV-specific outcomes will be based on the first positive laboratory-confirmed PCR test from a respiratory specimen during a healthcare encounter in a KPNC healthcare setting, occurring during the relevant follow-up window. RSV-positive test results will be combined with International Classification of Diseases, Tenth Revision, Clinical Modification (ICD-10-CM) diagnostic codes to define the RSV-specific outcomes. RSV-specific outcomes will include: PCR-confirmed RSV, PCR-confirmed RSV hospitalization, PCR-confirmed RSV LRTD, and PCR-confirmed RSV LRTD hospitalization.

Non-specific all-cause infant outcomes will include: all-cause LRTD, all-cause LRTD hospitalization, acute otitis media, and new antibiotic prescription (for any diagnosis). Identification of these outcomes will be based on ICD-10-CM diagnostic codes documented in infant EMRs during a healthcare encounter in a KPNC healthcare setting, occurring during the relevant follow-up window.

ELIGIBILITY:
Inclusion Criteria

Pregnant Individuals - Inclusion Criteria:

Participants must meet all of the following inclusion criteria to be eligible for inclusion in the study:

1. Gestational age at delivery ≥32 0/7 weeks of gestation (earliest gestational age eligible for ABRYSVO vaccination) during the study period
2. Maternal age 18 to 50 years at pregnancy onset
3. At least 1 prenatal visit between pregnancy onset and 20 weeks of gestation
4. Continuous KPNC enrollment for a minimum of 30 days prior to pregnancy onset through to the date of delivery, with no more than a 1-month administrative gap in coverage

Infants - Inclusion Criteria:

Participants must meet all of the following inclusion criteria to be eligible for inclusion in the study:

1. Born to a pregnant individual who has met all inclusion and exclusion criteria outlined above
2. Live birth
3. Enrolled as member in KPNC by 3 months of age

Exclusion Criteria

Pregnant Individuals - Exclusion Criteria:

Participants meeting any of the following criteria will not be included in the study:

1. Received any licensed or investigational RSV vaccine other than ABRYSVO at any time during pregnancy
2. Received ABRYSVO at ≥37 weeks' gestation
3. Received ABRYSVO at <32 0/7 weeks' gestation

Infants - Exclusion Criteria:

There are no exclusion criteria for infants. Those who receive any licensed or investigational RSV preventative product (e.g., monoclonal antibodies) at/after birth or any licensed or investigational RSV therapeutic (e.g., antiviral medications) will not be excluded, but their follow-up time will be censored on the date of receipt of the RSV preventative or therapeutic product.

Ages: 0 Years to 50 Years | Sex: All
Age Groups: Child, Adult
Study Population: The study population will comprise eligible maternal-infant pairs over a 2-year study period, identified from EMR records in the existing databases, which accrue in real-time as pregnancies/births occur. All pregnancies that reach 32 0/7 weeks' gestation during the 2-year study period, from September 22, 2023 (start of ABRYSVO vaccination season 1) to January 31, 2025 (estimated end of ABRYSVO vaccination season 2) will be eligible for inclusion, along with all live born infants from the eligible pregnancies. The KPNC pregnancy database will be used to identify the maternal-infant study population. This database links records of newborn infants with their mother, enabling integration of maternal data from across pregnancy and delivery encounters, along with infant birth information and longitudinal follow-up for infants who remain enrolled with KPNC. Infant healthcare encounters after the birth and throughout the follow-up period will be identified in the EMR.
Sampling Method: Non-Probability Sample
Enrollment: 39456 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Polymerase chain reaction (PCR)-confirmed RSV LRTD occurring ≤180 days after birth (first episode). | ≤180 days after birth
  To estimate VE of ABRYSVO vaccination during pregnancy against RSV LRTD among infants from birth through 6 months of age.

SECONDARY OUTCOMES:
Key Secondary 1: PCR-confirmed RSV LRTD hospitalization occurring ≤180 days after birth (first episode). | ≤180 days after birth
  To estimate VE of ABRYSVO vaccination during pregnancy against RSV LRTD hospitalization among infants from birth through 6 months of age.
Secondary 1: PCR-confirmed RSV occurring ≤180 days after birth (first episode). | ≤180 days after birth
  To estimate VE of ABRYSVO vaccination during pregnancy against RSV among infants from birth through 6 months of age.
Secondary 2: PCR-confirmed RSV hospitalization occurring ≤180 days after birth (first episode). | ≤180 days after birth
  To estimate VE against RSV hospitalization among infants from birth through 6 months of age.
Secondary 3: LRTD (any cause) occurring ≤180 days after birth (first episode during the RSV season). | ≤180 days after birth
  To estimate VE against all-cause LRTD among infants born in-season from birth through the RSV season (through 6 months of age).
Secondary 4: LRTD hospitalization (any cause) occurring ≤180 days after birth (first episode during the RSV season). | ≤180 days after birth
  To estimate VE against all-cause LRTD hospitalization among infants born in-season from birth through the RSV season (through 6 months of age).
Secondary 5: Acute otitis media occurring ≤180 days after birth (first episode during the RSV season). | ≤180 days after birth
  To estimate VE against acute otitis media among infants born in-season from birth through the RSV season (through 6 months of age).
Secondary 6: New antibiotic prescriptions occurring ≤180 days after birth (first prescription during the RSV season). | ≤180 days after birth
  To estimate VE against new antibiotic prescriptions among infants born in-season from birth through the RSV season (through 6 months of age).
Secondary 7: PCR-confirmed RSV occurring ≤360 days after birth (first episode). | ≤360 days after birth
  To estimate VE and interval-specific VE against RSV among infants from birth through 12 months of age.
Secondary 8: PCR-confirmed RSV hospitalization occurring ≤360 days after birth (first episode). | ≤360 days after birth
  To estimate VE and interval-specific VE against RSV hospitalization among infants from birth through 12 months of age.
Secondary 9: PCR-confirmed RSV LRTD occurring ≤360 days after birth (first episode). | ≤360 days after birth
  To estimate VE and interval-specific VE of ABRYSVO vaccination during pregnancy against RSV LRTD among infants from birth through 12 months of age.
Secondary 10: PCR-confirmed RSV LRTD hospitalization occurring ≤360 days after birth (first episode). | ≤360 days after birth
  To estimate VE and interval-specific VE of ABRYSVO vaccination during pregnancy against RSV LRTD hospitalization among infants from birth through 12 months of age.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3671048